CLINICAL TRIAL: NCT01220726
Title: Randomized Double-blind Placebo Controlled Trial of Intradetrusor Injections of Botox for the Treatment of Refractory Overactive Bladder Secondary to Benign Prostatic Obstruction-BTX0621
Brief Title: Botox for the Treatment of Overactive Bladder Secondary to Benign Prostatic Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTX0621
Record Dates: First submitted 2010-06-22; First posted 2010-10-14 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Overactive Bladder
Keywords: OAB
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Active Comparator): 200U onabotulinumtoxinA (botox)
  Interventions: Drug: Botox
- Placebo (Placebo Comparator): 200U Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botox — Botox injection
  Arms: Botox
Drug: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind study comparing intravesical injection of BOTOX to placebo. Study subjects will be randomized (1:1 ratio) to one of the following treatment groups:

DETAILED DESCRIPTION:
Group 1 n=20 BOTOX® 200U Group 2 n=20 Placebo BOTOX® (saline) At Visit 2 (Treatment, Day 0), subjects will receive one injection cycle of BOTOX (200U) or placebo (saline). The study duration is approximately 284 days and consists of a Screening Visit (Day -7 to -14), a Treatment/Randomization Visit (Visit 2, Day 0), and Follow-up Visits at 7, 30, 90, 180, and 270 Days. Telephone Follow-ups will be made 3 days following the injection cycle.

Subjects demonstrating an insufficient response to treatment may receive an open-label injection cycle of BOTOX (200U) at Day 90. Subjects receiving this injection will re-commence Follow-up Visits and be followed for an additional 270 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male outpatients of any race, between 40 and 90 years of age.
2. Clinical signs and symptoms of frequency (>=8 micturitions/day) and urgency (>=2 episodes/day).
3. Urodynamic history consistent with OAB that developed in conjunction with BPO and that persists for at least 3 months post TURP or PVP, RRP or other obstruction relieving procedure.
4. OAB inadequately controlled with anticholinergic medications, as per Investigator opinion.
5. Qmax >12mL/s with a voided volume of >125mL.
6. IPSS >12, with IPSS QoL >3 at study Visit 1.
7. Willing to use clean intermittent catheterization (CIC) to empty the bladder or is willing to have an indwelling catheter, if necessary following study treatment.
8. Able to understand the requirements of the study, including completing questionnaires and signing Informed Consent/HIPAA.

Exclusion Criteria:

1. Known history of interstitial cystitis, uninvestigated hematuria, bladder outlet obstruction due to vesical neck contracture, mullerian duct cysts, urethral obstruction due to stricture/valves/sclerosis of urethral tumor, radiation cystitis, genitourinary tuberculosis, bladder calculi, or detrusor-sphincter dyssynergia.
2. Known history of clinically significant cardiovascular disease, cerebrovascular disease, or arrhythmia.
3. History of spinal cord injury or multiple sclerosis, or other neurological disease which may be contributing to OAB.
4. Known history of hydronephrosis.
5. Current indwelling catheter, or removal of chronic catheter <1 month prior to study entry.
6. Non-compliance with wash-out periods for prohibited medications/therapies (Supplement I).
7. Evidence of Urinary Tract Infection according to local standard of care.
8. Serum PSA of >10ng/mL.
9. 24 hour total volume voided >3000 mL of urine. [As determined by completion of a patient bladder diary during the screening period]
10. Medical condition that may increase their risk of exposure to botulinum toxin including diagnosed Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
11. Allergy or sensitivity to any component of BOTOX® (Section 5.2).
12. Known uncontrolled systemic disease.
13. Evidence of recent alcohol/drug abuse.
14. Subjects who, in the opinion of the Investigator, have a significant condition that puts them at significant risk, may confound study results, or interfere with study participation.
15. History of poor cooperation, non-compliance with medical treatment, or unreliability.

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2012-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Te, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total number of participants recruited and enrolled was 30. A total of 28 completed the study.
Period: Overall Study
Arm/Group | Botox | Placebo
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox | Placebo | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Median (Full Range); unit: years] | 80 [48 to 87] | 68 [53 to 83] | 74 [48 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 13 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28
BMI [Median (Full Range); unit: kg/m^2] | 25.7 [20 to 30.4] | 32.5 [24 to 38] | 28 [20 to 38]
Baseline International Prostate Symptom Score [Median (Inter-Quartile Range); unit: units on a scale] — International Prostate Symptom Score (IPSS) is a 7 point scale used to screen, track and manage symptoms associated with BPH. The symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Scores range from 1 to 5 for a total of maximum 35 points (0-7 Mildly symptomatic, 8-19 Moderately symptomatic, 20-35 Severely symptomatic).
  units on a scale | 16 [13 to 23] | 20 [12 to 23] | 18 [12.5 to 23]
Baseline maximum flow rate (Qmax) [Mean (Standard Deviation); unit: mL/s] — Maximum flow rate (Qmax) is the the maximum recorded flow rate
  mL/s | 21.1 (10.5) | 16.0 (5.8) | 18.6 (8.15)
Baseline Voided Volume [Mean (Standard Deviation); unit: mL] — Voided volume is the amount of urine output during a micturition.
  mL | 265.4 (132.3) | 212.6 (74.5) | 239 (103.4)
Baseline postvoid residual volume (PVR) [Mean (Standard Deviation); unit: mL] — Postvoid residual volume (PVR) is the volume of fluid remaining in the bladder immediately after the completion of micturition.
  mL | 38.3 (39.5) | 34.8 (31.2) | 36.55 (35.35)
Baseline Voiding frequency [Median (Inter-Quartile Range); unit: times voided] — This is the frequency of micturitions during a 24-hour period.
  times voided | 11 [9 to 14] | 10.5 [8 to 13] | 10.75 [9 to 14]
Type of Procedure: TURP or Laser [Number; unit: participants] — Transurethral resection of the prostate (TURP) involves resecting the prostatic tissue, while a laser procedure involves vaporizing the tissue using a laser.
  participants
    TURP | 6 | 6 | 12
    Laser | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Urinary Frequency
Description: This is the measure of urinary frequency at baseline for those in the placebo and botox arms to day 270
Time Frame: From Baseline to Day 270
Measure: Median (Inter-Quartile Range); unit: urinations
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
urinations
  Baseline | 10.5 [8 to 13] | 11 [9 to 14]
  Day 7 | 12 [9 to 14] | 8.5 [7 to 12.5]
  Day 30 | 12 [8 to 13] | 8 [7 to 10]
  Day 90 | 13 [7 to 13] | 8 [7 to 12]
  Day 180 | 10 [8 to 14] | 9 [8 to 12]
  Day 270 | 8.5 [5 to 10] | 9.5 [7 to 10]

2. Primary Outcome: Urgency
Description: This measured the degree of urinary urgency using a 3-day voiding diary. Patients were assessed for the number of urgency episodes they had by answering yes or no.
Time Frame: From Baseline to Day 270
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
episodes
  Baseline | 4.5 [1 to 10] | 2 [2 to 4]
  Day 7 | 0.5 [0 to 3] | 1 [0 to 6]
  Day 30 | 0 [0 to 2] | 0 [0 to 1]
  Day 90 | 0 [0 to 1] | 0 [0 to 1]
  Day 180 | 1 [0 to 3] | 1.5 [0 to 4]
  Day 270 | 0 [0 to 1] | 0 [0 to 7]

3. Primary Outcome: Quality of Life (QoL)
Description: Quality of Life (QoL) is from the ICIQ-QAB (international Consultation of Incontinence Overactive Bladder) Questionnaire. It is scored 25-160 and those with higher scores have higher impact on quality of life.
Time Frame: From Baseline to Day 270
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
scores on a scale
  Baseline | 90 [79 to 93] | 73 [60 to 92]
  Day 7 | 97.5 [82.5 to 100.5] | 81.5 [47 to 92]
  Day 30 | 92 [90 to 94] | 82.5 [63 to 94]
  Day 90 | 91 [66 to 103] | 88 [61 to 91]
  Day 180 | 97.5 [88.5 to 105.5] | 79 [59 to 86]
  Day 270 | 99 [93 to 107] | 79 [67 to 87]

4. Primary Outcome: International Consultation on Incontinence Questionnaire (ICIQ)
Description: ICIQ is a brief validated instrument that is comprehensive for the assessment of incontinence and measures frequency, severity and impact on quality of life. There are a total of 23 items. The overall score ranges from 1-84 with greater values indicating increased symptom severity. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient.
Time Frame: From Baseline to Day 270
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
units on a scale
  Baseline | 7 [5 to 12] | 9 [4 to 15]
  Day 7 | 5 [3 to 7] | 8 [5 to 11]
  Day 30 | 4.5 [1 to 8] | 7 [5 to 10]
  Day 90 | NA [NA to NA] — Insufficient number of participants with this event. | NA [NA to NA] — Insufficient number of participants with this event.
  Day 180 | 4 [1 to 6] | 4 [4 to 7]
  Day 270 | 4 [3 to 4] | 8.5 [6 to 13]

5. Primary Outcome: Postvoid Residual Volume (PVR)
Description: Postvoid residual volume (PVR) is the volume of fluid remaining in the bladder immediately after the completion of micturition.
Time Frame: From Baseline to Day 270
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
mL
  Baseline | 34.8 (31.2) | 36 (39.5)
  Day 7 | 41.7 (NA) — After extensive research and review of files, standard deviation cannot be located. | 137.1 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 30 | 26.3 (NA) — After extensive research and review of files, standard deviation cannot be located. | 73.1 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 90 | NA (NA) — Insufficient number of participants with this event. | NA (NA) — Insufficient number of participants with this event.
  Day 180 | 151.6 (NA) — After extensive research and review of files, standard deviation cannot be located. | 168.6 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 270 | 21.2 (NA) — After extensive research and review of files, standard deviation cannot be located. | 54.4 (NA) — After extensive research and review of files, standard deviation cannot be located.

6. Primary Outcome: Maximum Flow Rate (Qmax)
Description: Qmax is the the maximum recorded flow rate
Time Frame: From Baseline to Day 270
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
mL/s
  Baseline | 16.0 (5.8) | 21.1 (10.5)
  Day 7 | 14 (NA) — After extensive research and review of files, standard deviation cannot be located. | 15.7 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 30 | 12.7 (NA) — After extensive research and review of files, standard deviation cannot be located. | 16.5 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 90 | 13.9 (NA) — After extensive research and review of files, standard deviation cannot be located. | 10.3 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 180 | 8.7 (NA) — After extensive research and review of files, standard deviation cannot be located. | 12.8 (NA) — After extensive research and review of files, standard deviation cannot be located.
  Day 270 | 9.3 (NA) — After extensive research and review of files, standard deviation cannot be located. | 12.9 (NA) — After extensive research and review of files, standard deviation cannot be located.

7. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: International Prostate Symptom Score (IPSS) -is a 7 point scale used to screen, track and manage symptoms associated with BPH. The symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Scores range from 1 to 5 for a total of maximum 35 points (0-7 Mildly symptomatic, 8-19 Moderately symptomatic, 20-35 Severely symptomatic)
Time Frame: From Baseline to Day 270
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Botox
Number analyzed (Participants) | 13 | 15
units on a scale
  Baseline | 20 [12 to 23] | 16 [13 to 23]
  Day 7 | 13.5 [8 to 20] | 15.5 [13 to 25]
  Day 30 | 13 [11 to 18] | 15 [8 to 18]
  Day 90 | 16 [10 to 24] | 10 [5 to 17]
  Day 180 | 14.5 [11 to 19.5] | 17 [13 to 22]
  Day 270 | 17 [10 to 18] | 15 [12 to 15]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over 1 year
Groups:
- Botox: Number of adverse events that occurred in the botox arm
- Placebo: Number of adverse events that occurred in the placebo arm
Arm/Group | Botox | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 4/15 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botox (N=15) | Placebo (N=13)
Hematuria (Renal and urinary disorders) | 1 | 0
Acute Urinary retention (Renal and urinary disorders) | 2 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No